CLINICAL TRIAL: NCT03850353
Title: Obstructive Sleep Apnea Syndrome (OSAS) and Dizziness
Acronym: OSASDiz
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0920-18-TLV
Record Dates: First submitted 2019-02-13; First posted 2019-02-21 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Sleep Apnea Syndromes, Obstructive; Dizziness; Eustachian Tube Dysfunction
MeSH Terms: conditions — Sleep Apnea Syndromes; Dizziness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- OSAS: Patients with Obstructive Sleep Apnea (AHI>15 in a sleep study)
- Dizziness: Patients with Dizziness (defined as a non-spinning sensation, without illusion of movement)
- No OSAS No Dizziness: Patients without dizziness and no evidence for OSAS (subjects referred for the ENT or the Sleep clinic with no dizziness and no evidence of OSAS )

SUMMARY:
A total of 400 participants will be recruited: 200 patients with suspected OSAS will be recruited from the sleep clinic (OSAS group), 100 patients diagnosed with dizziness will be recruited from the ENT clinic (Dizziness group). In addition, 100 patients with no dizziness and no evidence for OSAS will be recruited from both the sleep clinic and the ENT clinic (controls). Informed consents will be completed by all participants. ). In order to assess the effect of treatment of OSAS on dizziness -patients with the diagnosis of OSAS will complete validated questionnaires regarding sleep, dizziness and eustachian tube function 3 months following initiation of treatment with CPAP

DETAILED DESCRIPTION:
Group 1 - 200 patients with OSAS based on sleep study will be recruited from the sleep clinic (OSAS group) Group 2 - 100 patients diagnosed with dizziness will be recruited from the ENT clinic (Dizziness group).

Group 3 - 100 patients with no dizziness and no evidence for OSAS will be recruited from both the sleep clinic and the ENT clinic (controls).

Informed consents will be completed by all participants. All participants will undergo thorough physical examination with particular attention to the vestibular system, otoscopy, examination of the pharynx including with a flexible endoscope (that is part of the standard ENT examination). The examiner will photo-document the nasopharynx as needed.

Demographics and complete medical history will be recorded for each participant.

All participants will complete the following validated questionnaires:

1. Berlin questionnaire for OSAS
2. Epworth sleepiness scale
3. Dizziness Handicap Inventory - Hebrew version (DHI-H)
4. Eustachian tube dysfunction questionnaire Subjects from Group 1 that will have positive dizziness/eustachian dysfunction will be referred for the ENT clinic for further evaluation. Participants with dizziness will be treated, if indicated, based on their diagnosis and according to clinical guidelines with symptoms relievers in the acute phase (medications such sulpiride; fluids, metoclopramide) , physiotherapy and thiazide diuretics for chronic conditions.

Patients from Group 2 that will have a positive Berlin questionnaire will undergo ambulatory sleep study with WatchPAT (Itamar Medical, Israel). The Berlin questionnaire consists of 10 items divided into 3 categories (category 1: items 1-5, category 2: items 6-9, category 3: item 10). A positive Berlin question (high risk for OSA) is when 2 out of the 3 categories are positive.

A patient will be diagnosed with OSAS if the Apnea-Hypopnea Index in the sleep study will be greater than 5 per hour of sleep. Patients with moderate-severe OSA (AHI greater than 15 per hour of sleep) will be treated with CPAP.

Patients from Group 3 with positive Berlin questionnaire will be referred for a sleep study as indicated in the clinical setting.

Risk factors associated with OSAS will be recorded: Age, gender, smoking, BMI, neck circumference. In addition, comorbidities associated with OSAS will be recorded such as hypertension, diabetes, hyperlipidemia, coronary artery disease and stroke.

The investigators expect 15% of the patients referred to the sleep study to be diagnosed with OSAS.

In order to assess the effect of treatment of OSAS on dizziness -patients with dizziness and diagnosis of moderate severe OSAS (AHI >15) who will be treated with CPAP will be asked to complete the 4 validated questionnaires 3 months following initiation of treatment with CPAP. CPAP use of 80% or more of total sleep time (T.S.T) will be considered as full compliance. 60-80% of T.S.T- partial compliance. <60% - no compliance.

ELIGIBILITY:
Inclusion Criteria:

* age 18-90 years
* Group 1: subjects diagnosed with OSAS based sleep study
* Group 2: subjects referred to the ENT clinic with major complaint of dizziness (defined as a non-spinning sensation, without illusion of movement)
* Group 3: subjects referred for the ENT or the Sleep clinic with no dizziness and no evidence of OSAS

Exclusion Criteria:

* Neurological and psychiatric disorders
* Pregnant women
* Subjects with judgment difficulties
* Subjects that will be diagnosed with specific pathology that explains their dizziness.
* Subjects previously diagnosed and treated surgically for OSAS .
* Subjects with any previous intervention on the soft palate base tongue or pharynx (not including adenotonsillectomy).
* Subjects with any congenital anomaly of the palate and pharynx

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1 - 200 patients with OSAS based on sleep study will be recruited from the sleep clinic (OSAS group) Group 2 - 100 patients diagnosed with dizziness will be recruited from the ENT clinic (Dizziness group).
  Group 3 - 100 patients with no dizziness and no evidence for OSAS will be recruited from both the sleep clinic and the ENT clinic (controls).
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
The change in the score on Dizziness Handicap Inventory (DHI) | 3 months after beginning of use of CPAP
  The change in the total score on the DHI before and after the use of CPAP in (minimum score:0, maximum score: 100. Higher values represent worsening of the dizziness) OSAS patients